CLINICAL TRIAL: NCT04849039
Title: "Pulmonary Microbiota and Related Immunity Role in Predicting Ventilator Associated- Pneumonia (VAP) Development in Mechanical Ventilated Patients"
Brief Title: Lung Microbiota and VAP Development (PULMIVAP)
Acronym: PULMIVAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: San Gerardo Hospital (Other); University of Parma (Other)
Responsible Party: Sponsor
Other Study IDs: 1469-23.07.2019
Record Dates: First submitted 2021-02-24; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-02

CONDITIONS: Mechanical Ventilation
Keywords: Observational; Cohort Study; Ventilator-associated pneumonia; Mechanical Ventilation; Lung microbiota
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tracheal aspirate; Oropharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanicaly ventilated adult patients for non-pulmonary conditions

SUMMARY:
Ventilator-associated pneumonia (VAP) refers to a lower respiratory tract nosocomial infection acquired >48h after being intubated in Intensive Care Units. Pathogenesis of VAP is mechanical and associated with microaspiration and leakage of oropharyngeal secretions around the endotracheal tube. A novel approach to VAP will attempt to explore how the abrupt ecological order of acute infection (high bacterial biomass, low community diversity) emerges from the dynamic homeostasis of a pre-existing ecosystem in which lung microbiota and local immunity interaction play their essential role.

Therefore, the investigators aim to explore if oral and lung microbiota modifications with local immunity changes, contribute in the pathogenesis of VAP in patients intubated for non-pulmonary reasons. Early changes in the host microbiota with the innate immunity system impairs tissue homeostasis and may represent a new distinct condition and a potential tool for early diagnosis and prevention of VAP.

DETAILED DESCRIPTION:
Several factors are involved in the pathogenesis of VAP: the presence of endotracheal tube, the creation of bacterial biofilms around the device, host characteristics (comorbidities, surgery, antibiotic exposure) and, finally, immunological factors (including modulation of cytokine expression). In this study, patients mechanically ventilated for non-pulmonary reasons, will be followed up to 15 days of ventilation, estubation or death (whichever comes first). For microbiota analysis, all patients who develop VAP in the first 15 days of MV will be selected and matched (1:1; by center, gender, age (+/- 10 years), reason for intubation, duration of intubation), with a patient who do not developed VAP during MV. The optimal matching algorithm will be used to identify the control group that minimizes the total intra-pair dissimilarity.

The investigators plan to enroll about 700 MV patients for non-pulmonary conditions in order to describe VAP and non-VAP patients' characteristics identify. The investigators estimate that at least 70 patients will develop VAP in the first 15 days of MV. Microbiota and immunological analysis will be longitudinally performed on tracheal aspirate samples and oro-pharyngeal swab. The investigators will performe microbiota analyses on tracheal aspirate and oropharyngeal swab according to the following time schedule:

* VAP patient, 3 times: intubation (T0), the 24h before VAP development (T pre-VAP) and at VAP development (T-VAP).
* non-VAP patient, 2 times: intubation (T0) and a second sample, selected at the time point (day), corresponding to T-VAP of his/her matched VAP-patient (T no-VAP).

The investigators will perform immunological analysis on tracheal aspirate for all patients at intubation and at T-VAP or T no-VAP time.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Patients ventilated for reasons other than pulmonary failure with an expected need for MV longer than 48 hours

Exclusion Criteria:

* Admission in ICU with a pneumonia
* Clinical Pulmonary Infectious Score (CPIS) > 6
* Antibiotic therapy > 3 days prior to the start of MV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients mechanicaly ventilated for non pulmonary conditions
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Lung/oral microbiota and VAP development | (Time frame for VAP patients: intubation (T0), 24h before VAP development (T pre- VAP) and at VAP development (T-VAP). Time frame for non-VAP patients: intubation (T0), samples corresponding to T-VAP of matched VAP patients (T no VAP))
  Alfa and beta diversity variation based on 16S-rRNA sequencing in tracheal aspirates and oral samples.
  To explore the association between the composition and related changes over time of the lung/oral microbiota and VAP development has been used the measure of the alfa-diversity (number of different OTUs in each sample) and beta-diversity (similarity between samples in terms of OTUS composition).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico, Milan, MI, Italy

REFERENCES:
- [Background] Spalding MC, Cripps MW, Minshall CT. Ventilator-Associated Pneumonia: New Definitions. Crit Care Clin. 2017 Apr;33(2):277-292. doi: 10.1016/j.ccc.2016.12.009. Epub 2017 Jan 18. PMID 28284295
- [Background] Emonet S, Lazarevic V, Leemann Refondini C, Gaia N, Leo S, Girard M, Nocquet Boyer V, Wozniak H, Despres L, Renzi G, Mostaguir K, Dupuis Lozeron E, Schrenzel J, Pugin J. Identification of respiratory microbiota markers in ventilator-associated pneumonia. Intensive Care Med. 2019 Aug;45(8):1082-1092. doi: 10.1007/s00134-019-05660-8. Epub 2019 Jun 17. PMID 31209523
- [Background] Zakharkina T, Martin-Loeches I, Matamoros S, Povoa P, Torres A, Kastelijn JB, Hofstra JJ, de Wever B, de Jong M, Schultz MJ, Sterk PJ, Artigas A, Bos LDJ. The dynamics of the pulmonary microbiome during mechanical ventilation in the intensive care unit and the association with occurrence of pneumonia. Thorax. 2017 Sep;72(9):803-810. doi: 10.1136/thoraxjnl-2016-209158. Epub 2017 Jan 18. PMID 28100714
- [Background] Shimizu T, Kono M, Watanabe H, Adachi S, Hasegawa M, Okuda K, Tanaka K, Kameda K, Hirota S, Sako M. [CT evaluation in the diagnosis of pulmonary nodules using lung phantom]. Nihon Igaku Hoshasen Gakkai Zasshi. 1987 Oct 25;47(10):1251-9. No abstract available. Japanese. PMID 3441423
- [Background] Martin-Loeches I, Dickson R, Torres A, Hanberger H, Lipman J, Antonelli M, de Pascale G, Bozza F, Vincent JL, Murthy S, Bauer M, Marshall J, Cilloniz C, Bos LD. The importance of airway and lung microbiome in the critically ill. Crit Care. 2020 Aug 31;24(1):537. doi: 10.1186/s13054-020-03219-4. PMID 32867808
- [Background] Yatera K, Mukae H. Drastic change in the lung microbiome induced by mechanical ventilation. Respir Investig. 2020 Nov;58(6):425-426. doi: 10.1016/j.resinv.2020.07.005. Epub 2020 Sep 3. No abstract available. PMID 32893161
- [Background] Sommerstein R, Merz TM, Berger S, Kraemer JG, Marschall J, Hilty M. Patterns in the longitudinal oropharyngeal microbiome evolution related to ventilator-associated pneumonia. Antimicrob Resist Infect Control. 2019 May 22;8:81. doi: 10.1186/s13756-019-0530-6. eCollection 2019. PMID 31139364
- [Background] Dickson RP, Schultz MJ, van der Poll T, Schouten LR, Falkowski NR, Luth JE, Sjoding MW, Brown CA, Chanderraj R, Huffnagle GB, Bos LDJ; Biomarker Analysis in Septic ICU Patients (BASIC) Consortium. Lung Microbiota Predict Clinical Outcomes in Critically Ill Patients. Am J Respir Crit Care Med. 2020 Mar 1;201(5):555-563. doi: 10.1164/rccm.201907-1487OC. PMID 31973575
- [Background] Huebinger RM, Smith AD, Zhang Y, Monson NL, Ireland SJ, Barber RC, Kubasiak JC, Minshall CT, Minei JP, Wolf SE, Allen MS. Variations of the lung microbiome and immune response in mechanically ventilated surgical patients. PLoS One. 2018 Oct 24;13(10):e0205788. doi: 10.1371/journal.pone.0205788. eCollection 2018. PMID 30356313
- [Background] Yin Y, Hountras P, Wunderink RG. The microbiome in mechanically ventilated patients. Curr Opin Infect Dis. 2017 Apr;30(2):208-213. doi: 10.1097/QCO.0000000000000352. PMID 28067677